CLINICAL TRIAL: NCT04116164
Title: A Phase 0 Study to Assess the Safety and Biodistribution of a Novel Radiolabeled Antibody Targeting Human Kallikrein-2 (hk2) in Subjects With Metastatic Castration-resistant Prostate Cancer.
Brief Title: Safety and Targeting of Anti-hk2 Antibody in mCRPC
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: SpectronRX (Industry)
Collaborators: Invicro (Other); Janssen Research & Development, LLC (Industry); Tomopath Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GID5490
Record Dates: First submitted 2019-10-01; First posted 2019-10-04 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Castration-Resistant Prostatic Cancer; Metastatic Disease
Keywords: Radiolabeled antibody; Imaging
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: 3-6 patients will be studied in each of 3 sub-cohorts to determine the most favorable mass amount of h11B6 (2 mg, 10 mg, 20 mg). An additional 6 patients will be imaged at the most favorable mass amount to assess tumor targeting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dosimetry and targeting (Experimental): Three sub-cohorts in cohort 1 will receive one slow bolus IV injection of 2 mg 111In-DOTA-h11B6 with 0, 8 and 18 mg unlabeled h11B6 respectively.
  In cohort 2, up to 6 patients will receive a slow bolus IV injection of 2 mg 111In-DOTA_h11B6 with any unlabeled h11B6 as determined from cohort 1, and will be imaged at one time-point
  Interventions: Drug: 111In-DOTA-h11B6

INTERVENTIONS:
Drug: 111In-DOTA-h11B6 — 4-6 mCi 111In labeled to 2 mg DOTA-h11B6; 0, 8 or 18 mg additional h11B6.

SUMMARY:
This is an imaging trial, to develop h11B6 as a therapeutic radiopharmaceutical for men with mCRPC.

This imaging study will be conducted to confirm the safety and estimate the mass amount of antibody h11B6, and confirm in vivo tumor targeting of the antibody, using Indium-111 (111In) radiolabeled h11B6 in subjects with advanced prostate cancer. This study will also provide the dosimetric information crucial for Phase 1 therapy.

DETAILED DESCRIPTION:
It is the intent to develop h11B6 as a therapeutic radiopharmaceutical for men with mCRPC. This Phase 0 study will be conducted to confirm the safety, estimate the mass amount, and confirm in vivo tumor targeting of the antibody. This study will use Indium-111 (111In) radiolabeled h11B6 in subjects with mCRPC to image known sites of disease and identify a favorable mass amount of antibody for satisfactory tumor targeting with minimal/no accumulation off-target. In cohort 1, In-111 labeled h11B6 will remain fixed at 2 mg, and additional h11B6 will be added in 2 sub-cohorts (8 mg and 18 mg respectively); up to 6 patients may be entered into a sub-cohort. Additional patients (up to 6) will be studied once the most favorable mass and imaging time point have been established, to establish targeting of antibody to known disease.

This study will provide the dosimetric information crucial for Phase 1 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mCRPC will be eligible if they meet the following criteria:
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Castrate levels of testosterone (<50 ng/dL [1.74 nmol/L])
* Metastatic disease documented by imaging
* Documented progressive mCRPC with androgen involvement as defined by - Prostate Cancer Working Group 3
* Acceptable laboratory parameters
* At least 28 days since administration of any therapeutic radioactive isotope
* Able to tolerate the conditions required to perform imaging studies (e.g., lying flat for at least 1 hour).

Exclusion Criteria:

* Known hypersensitivity to proteins, or other allergic diathesis that, in the opinion of the investigator, makes an immune response to humanized antibody likely
* Radiotherapy or immunotherapy within 30 days, or single fraction of palliative radiotherapy within 14 days of administration of study agent
* Any condition that, in the opinion of the Investigator, would impair the subject's ability to comply with study procedures and required study visits
* Active, symptomatic, or untreated brain metastases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is being carried out in prostate cancer which afflicts only men.
Enrollment: 27 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Serum pharmacokinetics | 6 months
  Serum clearance kinetics of 111In-DOTA-h11B6, only in cohort 1, at each mass amount of antibody (2, 10, and 20 mg).
Radioactivity Biodistribution | 6 months
  Radioactivity residence times in liver, kidneys and tumor, only in cohort 1, at each mass amount of antibody (2, 10, and 20 mg).
Radioactivity accumulation in known tumor sites | 9 months
  Number of known metastatic lesions in which there is increased uptake of 111In, in both cohorts 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Morris, MD, Principal Investigator — Memorial Hospital for Cancer and Allied Diseases
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darson MF, Pacelli A, Roche P, Rittenhouse HG, Wolfert RL, Young CY, Klee GG, Tindall DJ, Bostwick DG. Human glandular kallikrein 2 (hK2) expression in prostatic intraepithelial neoplasia and adenocarcinoma: a novel prostate cancer marker. Urology. 1997 Jun;49(6):857-62. doi: 10.1016/s0090-4295(97)00108-8. PMID 9187691
- [Background] Thorek DL, Watson PA, Lee SG, Ku AT, Bournazos S, Braun K, Kim K, Sjostrom K, Doran MG, Lamminmaki U, Santos E, Veach D, Turkekul M, Casey E, Lewis JS, Abou DS, van Voss MR, Scardino PT, Strand SE, Alpaugh ML, Scher HI, Lilja H, Larson SM, Ulmert D. Internalization of secreted antigen-targeted antibodies by the neonatal Fc receptor for precision imaging of the androgen receptor axis. Sci Transl Med. 2016 Nov 30;8(367):367ra167. doi: 10.1126/scitranslmed.aaf2335. PMID 27903863
- [Background] Thorek DL, Evans MJ, Carlsson SV, Ulmert D, Lilja H. Prostate-specific kallikrein-related peptidases and their relation to prostate cancer biology and detection. Established relevance and emerging roles. Thromb Haemost. 2013 Sep;110(3):484-92. doi: 10.1160/TH13-04-0275. Epub 2013 Aug 1. PMID 23903407
- [Background] Vilhelmsson Timmermand O, Larsson E, Ulmert D, Tran TA, Strand S. Radioimmunotherapy of prostate cancer targeting human kallikrein-related peptidase 2. EJNMMI Res. 2016 Dec;6(1):27. doi: 10.1186/s13550-016-0181-z. Epub 2016 Mar 17. PMID 26983637
- [Background] McDevitt MR, Thorek DLJ, Hashimoto T, Gondo T, Veach DR, Sharma SK, Kalidindi TM, Abou DS, Watson PA, Beattie BJ, Timmermand OV, Strand SE, Lewis JS, Scardino PT, Scher HI, Lilja H, Larson SM, Ulmert D. Feed-forward alpha particle radiotherapy ablates androgen receptor-addicted prostate cancer. Nat Commun. 2018 Apr 24;9(1):1629. doi: 10.1038/s41467-018-04107-w. PMID 29691406